CLINICAL TRIAL: NCT02887378
Title: Protocol for Anatomopathologic Analysis of Biopsies Using Hot Clamps
Acronym: PincesChaude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PI2014_843_0003
Record Dates: First submitted 2016-08-02; First posted 2016-09-02 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Endoscopy
Keywords: bronchial biopsy

ARMS (2):
- hot clamps (Experimental): reusable hot biopsy forceps
  Interventions: Device: hot clamps
- normal clamps (Active Comparator): normal clamps
  Interventions: Device: normal clamps

INTERVENTIONS:
Device: hot clamps — reusable hot biopsy forceps
  Arms: hot clamps
Device: normal clamps
  Arms: normal clamps

SUMMARY:
A cross-over study of the impact of histologic results of bronchial biopsies performed using hot clamps compared to bronchial biopsies using standard clamps

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients with no known hemorrhage risk, with an indication of endobronchial biopsy
* Patients with no contra-indication for bronchial endoscopy
* Patients with or without endobronchial tumors
* Patients who have provided written informed consent
* Patients with health insurance coverage

Exclusion Criteria:

* Refusal to be examined
* Contraindication for electrocoagulation (Pacemaker or metallic endobronchial prosthesis)
* Pregnant women
* Patients unable to provide voluntary informed consent, under (tutelage) or guardianship, or unable to come to the center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
use of reusable hot biopsy forceps | 2 years
  To show that the use of hot clamps (thermocoagulating) for endobronchial analysis does not affect the anatomopathologic interpretation of biopsies under certain conditions (with varying in intensity of current).

CONTACTS AND LOCATIONS:
Overall Officials: Youcef DOUADI, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - Ch Saint Quentin, Saint-Quentin